CLINICAL TRIAL: NCT02115152
Title: Phase II Neoadjuvant Trial of Capecitabine, Cyclophosphamide and Epirubicin for Patients With Axillary Lymph Node Positive Stage II-III Operable Breast Cancer
Brief Title: Neoadjuvant Trial of Capecitabine for Axillary Lymph Node Positive Operable Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jianlun Liu, Director of Department of Breast Surgery, Guangxi Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JLiu
Record Dates: First submitted 2014-03-24; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Capecitabine; Neoadjuvant therapy; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Capecitabine; Cyclophosphamide; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FEC (Active Comparator): Patients will be randomized to received 4 cycles of fluorouracil, epirubicin and cyclophosphamide before surgery, and 4 cycles of docetaxel after surgery.
  Interventions: Drug: fluorouracil; Drug: cyclophosphamide; Drug: Epirubicin
- XEC (Experimental): Patients will be randomized to received 4 cycles of capecitabine, epirubicin and cyclophosphamide before surgery, and 4 cycles of docetaxel and capecitabine after surgery.
  Interventions: Drug: capecitabine; Drug: cyclophosphamide; Drug: Epirubicin

INTERVENTIONS:
Drug: fluorouracil
  Arms: FEC
Drug: capecitabine
  Arms: XEC
Drug: cyclophosphamide
Drug: Epirubicin

SUMMARY:
This randomized phase II trial compared pathologic response rates (pCR) of early breast cancer following neoadjuvant fluorouracil-epirubicin-cyclophosphamide(FEC) and capecitabine-epirubicin-cyclophosphamide (XEC).

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-70 with histologically proven, core-biopsied, Stage II-III invasive breast cancer
* No distant disease

Exclusion Criteria:

- Inadequate heart or liver or kidney function

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
pathologic response rates (pCR) | The breast sample will be evaluaed on the day of surgery during the cycle 4, an expected average of 12 weeks.
  The absence of invasive tumor in the final surgical breast sample (stage yT0 or ypTis)

SECONDARY OUTCOMES:
DFS(Disease free survial) | Participants will be evaluated on Day 1 of each cycle during chemotherapy, and Day 1 every 3 months after completion of chemotherapy. The expected average of 5 years.
  Time from randmization to breast-cancer recurrence, or a second primay cancer(ecluding contralateral ducal carcinoma in situ), or death from any cause, whichever comes first
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Hematologic, renal, and hepatic funcion will be assessed after each cycle and at the end of therapy, an expected average of 3 weeks.
  Adverse events are classified accoding NCI CTC criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jianlun Liu, MD, Principal Investigator — Guangxi Medical University Cancer Center
Locations (1):
- Breast Cancer Surgery Department of Guangxi Medical University Cancer Center, Nanning, Guangxi, China